CLINICAL TRIAL: NCT05582356
Title: Effect of Preoperative Oral Carbohydrate Loading on Elderly Patient Quality of Recovery in Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Effect of Preoperative Oral Carbohydrate Loading on Elderly Patient Quality of Recovery in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-2023/06
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-03

CONDITIONS: Quality Of Recovery
Keywords: Oral Carbohydrate; Elderly Patient; Mini Mental State Examination
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate group (Group OC) (Experimental): Preoperative education will be provided by researchers to the patients on the ward before fluid intake. Solid food will be forbidden starting at 20:00 p.m, and drinking will be forbidden after 22:00 p.m the day before surgery. Group OC will consume carbohydrate fluid at 22.00 p.m. and two hours before the surgery
  Interventions: Dietary Supplement: Carbohydrate group (Group OC)
- Placebo group (Group OP) (Sham Comparator): Preoperative education will be provided by researchers to the patients on the ward before fluid intake. Solid food will be forbidden starting at 20:00 p.m, and drinking will be forbidden after 22:00 p.m the day before surgery. Group OP will consume an equal amount of water 22:00 p.m. and two hours before the surgery.
  Interventions: Dietary Supplement: Placebo group (Group OP

INTERVENTIONS:
Dietary Supplement: Carbohydrate group (Group OC) — Carbohydrate group (Group OC)
  Arms: Carbohydrate group (Group OC)
Dietary Supplement: Placebo group (Group OP — Placebo group (Group OP
  Arms: Placebo group (Group OP)

SUMMARY:
This prospective randomized controlled study will be aimed to evaluate the effect of preoperative oral carbohydrate loading on the elderly patient's quality of recovery and satisfaction in undergoing knee arthroplasty (TKA) surgery with spinal anesthesia.

DETAILED DESCRIPTION:
As an essential aspect of enhanced recovery after surgery, the advantages of preoperative oral carbohydrate loading (eg, improving patients' comfort during preoperative preparation, reducing nausea and vomiting, and reducing insulin resistance) have been shown by a large number of studies.

This study will be conducted as a single-center, prospective, randomized, double-blinded trial in a university hospital. Elderly ( > 65) patients scheduled for elective TKA will be screened for enrollment in the study. Patients will be randomized into an oral carbohydrate group (Group OC), and an oral placebo group (Group OP). Solid food will be forbidden starting at 20:00, and drinking will be banned after 22:00 the day before surgery. Oral carbohydrate preload will be administered to the Group OC. In Group OP, the blinded researcher will give an equal volume of placebo fluid orally at 22:00 and 2 hours before the operation in the ward. The participant will record that the liquid has been completely consumed

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to the American Society of Anesthesiologists (ASA) I-III
* Patients scheduled for total knee arthroplasty

Exclusion Criteria:

* Previous operation on same knee
* Hepatic or renal insufficiency
* Younger than 65 years old
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* ASA IV
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months, or daily oral morphine equivalent of >5mg/day for one month)
* impaired gastrointestinal motility
* Fasting glucose >200
* Acquired immunodeficiency
* Severe malnutrition

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-15 score | Postoperative 24th hour
  Minimum value: 0, Maximum value: 150, higher scores mean better.

SECONDARY OUTCOMES:
Quality of Recovery-15 score | preoperative, postoperative day 7
  Minimum value: 0, Maximum value: 150, higher scores mean better.
Numerical Rating Scale | 24 hours
  Range 0-10, 0=no pain, 10=the worse pain ever.
Opioid consumption | 24 hours
  Opioid consumption
Range of knee motion | 48 hours
  Range of knee motion
Patient mobilization | 48 hours
  Patient reporting time of first standing to the side of the bed and time up and go test 2 days
Patient well-being (thirst, hunger, mouth dryness, nausea and vomiting, fatigue) will be assessed just before the operating room admission | preoperative
  5: very satisfied, 4: somewhat satisfied, 3: neutral, 2: somewhat dissatisfied, 1: very dissatisfied
Mini Mental State Examination | preoperative and postoperatve day 1
  Mini Mental State Examination Scale (This scale is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.)
Sleep Quality measured with Likert Scale | One week after surgery
  Patients' perceived sleep quality will be assessed with a Likert scale. Likert scale is scored from Likert scale where 1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied and 5 = very satisfied
Glucose measurement | Postoperative 24th hour
  Glucose measurement

CONTACTS AND LOCATIONS:
Overall Officials: Betül Başaran, MD,DESA, Study Director — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)